CLINICAL TRIAL: NCT01265862
Title: Comparison of LMA-Fastrach® and I-gel® for Tracheal Intubation: Does the Use of the GlideRite® Endotracheal Tube in Combination With the I-gel® Improve Success Rate?
Brief Title: Does the Use of the GlideRite® Endotracheal Tube in Combination With the I-gel® Improve Intubation Success Rate?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NM2011-001
Record Dates: First submitted 2010-12-21; First posted 2010-12-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Intubation; General Anesthesia
Keywords: Tracheal intubation; Supraglottic airway devices; Patients undergoing general anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LMA-Fastrach® and GlideRite® tube (Active Comparator): * Induction of general anesthesia with 1,5-2,5 mg/kg propofol and 1-3 mcg/kg fentanyl and neuromuscular relaxation with 0,6 mg/kg of rocuronium.
  * Direct laryngoscopy, evaluation of laryngeal view grade according to Cormack-Lehane classification
  * Insertion of LMA-Fastrach®, establishment of ventilation
  * Evaluation of glottic view through LMA-Fastrach® using fibrescope
  * Tracheal intubation with the GlideRite® tube through the LMA-Fastrach®
  * With the endotracheal tube in place, the anaesthesiologist will proceed to the removal of supraglottic device
  Interventions: Procedure: Tracheal intubation through LMA-Fastrach®
- I-gel® and GlideRite® tube (Experimental): * Induction of general anesthesia with 1,5-2,5 mg/kg propofol and 1-3 mcg/kg fentanyl and neuromuscular relaxation with 0,6 mg/kg of rocuronium.
  * Direct laryngoscopy, evaluation of laryngeal view grade according to Cormack-Lehane classification
  * Insertion of I-gel®, establishment of ventilation
  * Evaluation of glottic view through I-gel® using fibrescope
  * Tracheal intubation with the GlideRite® endotracheal tube through the I-gel®
  * With the endotracheal tube in place, the anaesthesiologist will proceed to the removal of supraglottic device
  Interventions: Procedure: Tracheal intubation through I-gel®

INTERVENTIONS:
Procedure: Tracheal intubation through LMA-Fastrach® — Tracheal intubation through a supraglottic airway device (LMA-Fastrach®) using a GlideRite® endotracheal tube
  Arms: LMA-Fastrach® and GlideRite® tube
Procedure: Tracheal intubation through I-gel® — Tracheal intubation through a supraglottic airway device (I-gel®) using a GlideRite® endotracheal tube
  Arms: I-gel® and GlideRite® tube

SUMMARY:
The investigators aim to compare two different types of supraglottic devices for tracheal intubation in patients undergoing elective surgery under general anesthesia.

The investigators hypothesis is that the use of the I-gel® supraglottic airway device associated with a GlideRite® endotracheal tube will result in an equal success rate of fiberoptic tracheal intubation when compared to the LMA-Fastrach® associated with a GlideRite® endotracheal tube. Time to intubate with the I-gel® device should also be shorter.

DETAILED DESCRIPTION:
Supraglottic airway devices such as LMA-Fastrach® and I-gel® provide patent airways during general anesthesia.

The LMA-Fastrach® is designed to provide a conduit for blind or fiberscopically guided tracheal intubations. However, the success rate of tracheal intubation on the first attempt through this device varies between 50 and 87%.

The I-gel® is a newer device for airway management which, with its wide bore, allows direct passage of a tracheal tube. Recent studies suggest that the I-gel® is easy to insert and that limited experience is needed before a high success insertion rate is obtained. A recent study conducted in our center compared the LMA-Fastrach® to the I-gel® supraglottic airway device. Our results showed a lower success intubation rate in the I-gel® group. We noticed that there was a tendency for the endotracheal tube to impinge on the posterior and lateral aspect of the larynx. The endotracheal tube used for intubation in our study was a standard polyvinyl chloride (PVC) tube. We believe that an endotracheal tube with a flexible tip(GlideRite®) would increase the intubation success rate through the I-gel® device. However, based on our clinical experience with the GlideRite® tube, blind tracheal intubation through the I-gel® airway device may be associated with a low success rate related to a lack of rigidity of its tip. Its use in combination with a fibrescope could compensate for this weakness. A recent study performed on mannequins showed a comparable success intubation rate of 99% for the I-gel® and LMA-Fastrach® when associated to a fibrescope.

In this prospective randomized study, we will compare the performance of the LMA-Fastrach® and the I-gel® associated with a GlideRite® endotracheal tube for fiberoptic tracheal intubation in patients undergoing elective surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Patients undergoing elective surgery under general anesthesia, requiring endotracheal intubation

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) classification ≥ 4
* Contraindications to muscle relaxation
* Mouth opening less than 2 cm
* Patients at increased risk of regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
First attempt success rate of tracheal intubation | After successful insertion of tracheal tube before the beginning of surgery

SECONDARY OUTCOMES:
Time needed for successful insertion of a supraglottic device | After insertion of the device before the beginning of surgery
Time needed to obtain successful tracheal intubation | After tracheal intubation before the beginning of surgery
First attempt success rate of supraglottic device insertion | After insertion of the device before the beginning of surgery
Global success rate of supraglottic device insertion | After insertion of the device before the beginning of surgery
Fibreoptic view following the supraglottic device insertion | After insertion of the device before surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Massicotte, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada